CLINICAL TRIAL: NCT00006473
Title: A Phase II Study of Oxaliplatin in Relapsed and Refractory Non-Hodgkin's Lymphoma
Brief Title: Oxaliplatin in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02363; ID99-406; CDR0000068297 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-11-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Angioimmunoblastic T-cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Oxaliplatin

ARMS (1):
- Treatment (oxaliplatin) (Experimental): Patients receive oxaliplatin IV over 2 hours on day 1. Treatment repeats every 21 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP

SUMMARY:
Phase II trial to study the effectiveness of oxaliplatin in treating patients who have relapsed or refractory non-Hodgkin's lymphoma. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate to oxaliplatin in patients with relapsed or refractory non-Hodgkin's lymphoma.

II. Determine the treatment-related toxicity of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to histologic subtype (indolent vs aggressive).

Patients receive oxaliplatin IV over 2 hours on day 1. Treatment repeats every 21 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A maximum of 72 patients will be accrued for this study within 2-3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent or refractory non-Hodgkin's lymphoma (NHL) of any histologic subtype

  * Indolent

    * Follicular small cleaved cell
    * Follicular mixed cell
    * Small lymphocytic
    * Mucosa-associated lymphoid tissue (MALT)
    * Monocytoid B-cell
    * Waldenstrom's macroglobulinemia
  * Aggressive

    * Follicular large cell
    * Diffuse large cell
    * Immunoblastic
    * Mantle cell
    * Ki-1+ NHL
    * Peripheral T-cell
    * Angiocentric and angioimmunoblastic
    * Transformed lymphoma
* Bidimensionally measurable disease
* No more than 3 prior treatment regimens as follows:

  * Primary radiotherapy is 1 regimen
  * Combined therapy with radiotherapy and chemotherapy is 1 regimen
  * Alternating therapy is 1 regimen
* No known brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 50-100%
* WBC count at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* SGOT/SGPT no greater than 2.5 times upper limit of normal
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No neuropathy greater than grade 1
* No history of allergy to platinum compounds or antiemetics
* No uncontrolled illness
* No active infection
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No concurrent colony-stimulating factors during first course of therapy
* At least 4 weeks since prior chemotherapy
* At least 4 weeks since prior radiotherapy
* No other concurrent investigational drugs
* No concurrent antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2000-09; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 6 years
  Using a Simon's two-stage model.

SECONDARY OUTCOMES:
Duration of response | Up to 6 years
  Analyzed using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Anas Younes, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States